CLINICAL TRIAL: NCT03973372
Title: Advancing Liver Therapeutic Approaches (ALTA). The ALTA Consortium Study Group for the Management of Portal Hypertension - A 5-year Longitudinal Observational Study of Patients Undergoing Transjugular Intrahepatic Portosystemic Shunt (TIPS) Placement
Brief Title: ALTA TIPS: A 5-year Longitudinal Observational Study of Patients Undergoing TIPS Placement
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of California, San Francisco (Other); Scripps Health (Other); University of Wisconsin, Madison (Other); University of Florida (Other); University of Arizona (Other); Stanford University (Other); Columbia University (Other); Weill Medical College of Cornell University (Other); Baylor Scott and White Health (Other); Mayo Clinic (Other); University of Chicago (Other); W.L.Gore & Associates (Industry); University of Minnesota (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Lisa VanWagner, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU00208288
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cirrhosis, Liver; Transjugular Intrahepatic Portosystemic Shunt (TIPS)
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Baseline serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ALTA is a multicenter consortium focused on the management of portal hypertension. ALTA TIPS is a longitudinal observational study of patients who are undergoing transjugular intrahepatic portosystemic shunt (TIPS) placement. ALTA will create a database that will provide clinical parameters and outcomes of patients undergoing TIPS as part of their standard of care in hopes of answering key clinical questions.

DETAILED DESCRIPTION:
This is a 5-year prospective, longitudinal, observational study of all patients undergoing TIPS placement. The study will accrue patients until the goal of 1,000 subjects is reached. Subjects will be followed prospectively for up to a total of 5 years. Patients will be clinically managed by their local physicians per standard of care and no specific treatments or interventions will be dictated by their enrollment in this study. Patients will be consented to enroll in the study prior to TIPS placement or within 14 days after TIPS placement (such as in the event of emergent TIPS) and their pertinent clinical information will be then collected. Subjects may be consented electronically using REDCap eConsent or docusign. Pre-TIPS participants will be asked to complete a short set of questionnaires and one verbal assessment both pre-TIPS and post-TIPS during regularly scheduled visits with their treating hepatologist. Blood and rectal samples will be collected as optional procedures, and participation in these procedures will not affect participation in the study. Patients will be asked to consent to three different 5mL blood samples (total 15mL) at the time of TIPS from the peripheral, central, and portal venous circulation. A 5 ml peripheral sample will also be collected at months 1, 6, and 12 post-TIPS. The peripheral blood samples will occur either prior to TIPS (time 0) in the IR suite or at months 1, 6 and 12 post-TIPS. The central and portal venous blood sample will occur during the TIPS procedure in the IR suite. The total blood volume collection throughout the study will be 30mL. The rectal swab will be performed by the IR/ anesthesia team prior to the TIPS procedure in the IR suite. During the prospective post-TIPS period all medical records will be reviewed including clinical notes, laboratory values, radiographic results and medication changes and this data will be inputted into the database. Participants will be asked to also complete the same questionnaires regarding their quality of life and patient reported outcomes at prespecified timepoints post-TIPS, at a minimum 3 months and 12 months post-TIPS placement and then yearly thereafter. The hepatic encephalopathy assessments and AUDIT-C questionnaire will be conducted at month 1, 3, 6,12 and then yearly thereafter as part of their usual post-TIPS care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 able to provide consent or have a legally authorized consent in the event the subject is unable to consent due to a transient clinical condition
* Subject scheduled to undergo a TIPS procedure

Exclusion Criteria:

* Minors under the age of 18 at the time of enrollment
* Prisoners
* Pregnant Women
* Subjects undergoing TIPS placement as part of an investigational study outside of usual clinical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expect about 1000 people in the entire study nationally. The study population will consist of patients over the age of 18 undergoing a TIPS procedure.
Sampling Method: Non-Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To prospectively collect clinical information on the use and outcomes associated with contemporary real-world practice of Transjugular Intrahepatic Portosystemic Shunts (TIPS) | up to 5 years
  Transjugular Intrahepatic Portosystemic Shunt (TIPS) was first developed as a salvage tool for life threatening variceal bleeding or for the management of severe ascites refractory to medical therapy. Over the past decade there have been improvements in TIPS stent technology resulting in reduction in stent occlusions as well as increased experience of TIPS use. This increase in TIPS use has been paralleled by the expansion of indications for TIPS placement. As TIPS use has increased, so have the clinical questions surrounding the ideal conditions in which to successfully manage the indication for the procedure, while minimizing the unintended consequences of TIPS.
The goals of the ALTA consortium are to answer key clinical questions related to contemporary patterns of TIPS usage as well as clinical outcomes. | up to 5 years
  Recent data supports the use of TIPS for the early treatment of variceal bleeding, treatment of portal vein thrombus to permit successful liver transplantation and decompression of portal hypertension before planned abdominal surgery. Questions on TIPS use still remain. For example, what is the ideal stent diameter and degree of portal gradient pressure reduction required to optimally manage ascites or varices while minimizing hepatic decompensation and hepatic encephalopathy?
Create a database that will serve to inform and answer clinically related questions about the optimization of TIPS and management. | up to 5 years
  Currently, the major short-term complications related to TIPS are exacerbation of underlying cardiopulmonary issues and hepatic decompensation. The long-term complication, however, is hepatic encephalopathy which can often have a significant burden on quality of life and may result in additional procedures for constrainment or complete occlusion of the TIPS in severe cases. Although clinical outcomes of TIPS have been published, many of these reports are limited to single center sites with small sample sizes.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa VanWagner, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (14):
- United States (14):
  - University of Arizona, Phoenix, Arizona
  - Stanford, Redwood City, California
  - Scripps Health, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Northwestern, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University, New York, New York
  - Weill Cornell, New York, New York
  - Baylor Scott & White Liver Consultants of Texas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bommena S, Mahmud N, Boike JR, Thornburg BG, Kolli KP, Lai JC, German M, Morelli G, Spengler E, Said A, Desai AP, Junna S, Paul S, Frenette C, Verna EC, Goel A, Gregory D, Padilla C, VanWagner LB, Fallon MB; Advancing Liver Therapeutic Approaches (ALTA) Study Group. The impact of right atrial pressure on outcomes in patients undergoing TIPS, an ALTA group study. Hepatology. 2023 Jun 1;77(6):2041-2051. doi: 10.1097/HEP.0000000000000283. Epub 2023 Jan 19. PMID 36651170
- [Background] Boike JR, Thornburg BG, Asrani SK, Fallon MB, Fortune BE, Izzy MJ, Verna EC, Abraldes JG, Allegretti AS, Bajaj JS, Biggins SW, Darcy MD, Farr MA, Farsad K, Garcia-Tsao G, Hall SA, Jadlowiec CC, Krowka MJ, Laberge J, Lee EW, Mulligan DC, Nadim MK, Northup PG, Salem R, Shatzel JJ, Shaw CJ, Simonetto DA, Susman J, Kolli KP, VanWagner LB; Advancing Liver Therapeutic Approaches (ALTA) Consortium. North American Practice-Based Recommendations for Transjugular Intrahepatic Portosystemic Shunts in Portal Hypertension. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1636-1662.e36. doi: 10.1016/j.cgh.2021.07.018. Epub 2021 Jul 15. PMID 34274511
- [Background] Boike JR, Mazumder NR, Kolli KP, Ge J, German M, Jest N, Morelli G, Spengler E, Said A, Lai JC, Desai AP, Couri T, Paul S, Frenette C, Verna EC, Rahim U, Goel A, Gregory D, Thornburg B, VanWagner LB; Advancing Liver Therapeutic Approaches (ALTA) Study Group. Outcomes After TIPS for Ascites and Variceal Bleeding in a Contemporary Era-An ALTA Group Study. Am J Gastroenterol. 2021 Oct 1;116(10):2079-2088. doi: 10.14309/ajg.0000000000001357. PMID 34158464
- [Background] Ge J, Lai JC, Boike JR, German M, Jest N, Morelli G, Spengler E, Said A, Lee A, Hristov A, Desai AP, Junna S, Pokhrel B, Couri T, Paul S, Frenette C, Christian-Miller N, Laurito M, Verna EC, Rahim U, Goel A, Das A, Pine S, Gregory D, VanWagner LB, Kolli KP; Advancing Liver Therapeutic Approaches (ALTA) Study Group. Nonalcoholic Fatty Liver Disease and Diabetes Mellitus Are Associated With Post-Transjugular Intrahepatic Portosystemic Shunt Renal Dysfunction: An Advancing Liver Therapeutic Approaches Group Study. Liver Transpl. 2021 Feb;27(3):329-340. doi: 10.1002/lt.25949. Epub 2021 Jan 2. PMID 33217178
- [Background] Kwong AJ, Devuni D, Wang C, Boike J, Jo J, VanWagner L, Serper M, Jones L, Sharma R, Verna EC, Shor J, German MN, Hristov A, Lee A, Spengler E, Koteish AA, Sehmbey G, Seetharam A, John N, Patel Y, Kappus MR, Couri T, Paul S, Salgia RJ, Nhu Q, Frenette CT, Lai JC, Goel A; Re-Evaluating Age Limits in Transplantation (REALT) Consortium. Outcomes of Liver Transplantation Among Older Recipients With Nonalcoholic Steatohepatitis in a Large Multicenter US Cohort: the Re-Evaluating Age Limits in Transplantation Consortium. Liver Transpl. 2020 Nov;26(11):1492-1503. doi: 10.1002/lt.25863. Epub 2020 Oct 13. PMID 33047893

DOCUMENTS (1):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03973372/Prot_000.pdf